## The study took place on may 17<sup>th</sup> 2022. The observation period ended on may 20<sup>th</sup> 2022.

### **Preliminary Results – at 547 catheters in 537 Patients:**

Total: 537 Patients = 100 %
 Male 324 = 60.3%
 Female 213 = 39.7%

#### Distribution in access sites and sides:

- Internal Jugular Vein 449 = 82.1 %
  - o RIJV 378 = 84.2% 69.1 %
  - o LIJV 71 = 15.8% 13.0 %
- Subclavian Vein 63 = 11.5 %
  - o RSV 28 = 44.4% 5.1 %
  - o LSV 35 = 55.6% 6.4 %
- Femoral Vein 32 = 5.9 %
  - o RFV 17 = 53.1% 3.1 %
  - o LFV 15 = 46.9% 2.8 %
- Basilica 1 = 0.17 %
- External Jugular Vein 2 = 0.33 %

#### Types of central venous catheters used:

- Multiple Lumen CVC 416 = 77.8 %
- High Flow CVC 67 = 12.5 %
- Introducer Sheath 45 = 8.4 %
- Other 7 = 1.3 %

#### Ultrasound guidance (%) in central venous access procedures:

• **US guidance** 446 = 81.5 %

### Percentage of patients getting a central line

• On ventilator 337 = 61.6 %

# $\textbf{Malpositions} \text{ (here, introducer sheathes were not counted as well as two RA positions in neurosurgical patients being operated on the state of the state o$

in sitting positions) 30/490 = 6.1 %

| • | Right atrium (RA) | 20 |
|---|-----------------------------------------|----|
| • | Ipsilateral subclavian vein | 3 |
| • | Contralateral internal jugular vein | 1 |
| • | Ipsilateral brachiocephalic vein | 1 |
| • | Contralateral brachiocephalic vein | 1 |
| • | CVC reverted with U turn (US diagnosed) | 1 |
| • | Lumbal vein | 1 |
| • | Intrapleural position | 1 |
| • | Right axillar vein (ipsilateral) | 1 |

## Mechanical complications referred to 547 central venous access procedures:

#### 63/547 = 11.5 %

| • | Arterial cannulation | 2 |
|---|---------------------------------------------------------|---------|
| • | Failure (Abandonment of procedure at the intended site) | |
| • | Arrhythmia | 9 |
| • | Multiple punctures (≥ 3 skin punctu | res) 32 |
| | <ul> <li>Examples with failure to adva</li> </ul> | nce GW |
| | ■ LIJV | 2 |
| | ■ RSV | 2 |
| | ■ RIJV | 2 |
| • | Arterial punctures | 4 |
| • | Change of puncture site | 8 |
| • | Intrapleural position | 1 |
| • | Pneumothorax | 1 |
| • | Infusothorax | 1 |
| • | Hematoma local | 1 |
| • | Thrombosis 24 h after CVAP via RIJV | 1 |